CLINICAL TRIAL: NCT01650714
Title: Endoscopic Full Thickness Biopsy of the Gastric Wall in Patients With Refractory Idiopathic Gastroparesis: Pilot Study to Detect Neuromuscular and Immune Pathologic Changes
Brief Title: Endoscopic Full Thickness Biopsy, Gastric Wall.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elizabeth Rajan, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-000714
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Full thickness gastric biopsy (Experimental): Full thickness gastric biopsy
  Interventions: Other: Full thickness gastric biopsy; Procedure: Full thickness gastric biopsy

INTERVENTIONS:
Other: Full thickness gastric biopsy
Procedure: Full thickness gastric biopsy

SUMMARY:
The proposed study will assess the efficacy and safety of the innovative endoscopic technique for the acquisition of full thickness gastric muscle wall biopsies. Having access to full thickness biopsies will allow an increased understanding of the pathophysiology of gastrointestinal diseases such as functional gastrointestinal disorders, gastroparesis, pseudoobstruction and other motility disorders. This information is essential to development of more targeted and effective therapy than currently available. Despite the high prevalence of functional gastrointestinal disorders and its significant impact on social and health care costs, the underlying cause is not well understood and there is no effective specific treatment to successfully alleviate patient symptoms.

DETAILED DESCRIPTION:
Our group has studied a new endoscopic method using a submucosal endoscopy with mucosal flap (SEMF) technique to acquire full thickness gastric tissues successfully and safely in preclinical studies.

The proposed study will assess the efficacy and safety of the innovative endoscopic technique for the acquisition of full thickness gastric muscle wall biopsies. Having access to full thickness biopsies will allow an increased understanding of the pathophysiology of gastrointestinal diseases such as functional gastrointestinal disorders, gastroparesis, pseudoobstruction and other motility disorders. This information is essential to development of more targeted and effective therapy than currently available. Despite the high prevalence of functional gastrointestinal disorders and its significant impact on social and health care costs, the underlying cause is not well understood and there is no effective specific treatment to successfully alleviate patient symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic refractory idiopathic gastroparesis:

   1. The refractory nature of symptoms (e.g. based on nutritional failure, consideration for enteral or parenteral nutrition) will be determined by the physician/gastroenterologist who is the primary care provider for the patient's gastroparesis.
   2. Patients will have documentation within the last 2 years of delayed gastric emptying with >30% retained gastric contents at 4 hours based on 296 kcal solid-liquid, fat-containing standard meal gastric emptying test.
   3. The patient's physician will determine if this procedure may potentially provide prognostic and therapeutic options.
2. Age > 18 and < 70 years old
3. Hemoglobin (Hb) > 10g, platelets >150,000 and prothrombin time- international normalized ratio (INR) <1.5
4. Ability to give informed consent

Exclusion Criteria:

1. Prior oropharyngeal, esophageal, gastric or small bowel surgery
2. Esophageal stricture
3. Prior abdominal radiation therapy
4. Prior feeding tube placement
5. Coagulopathy
6. Use of Coumadin or anti-platelet drugs e.g. Plavix, steroids or immunosuppressive drugs
7. Pregnancy -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with successful endoscopic full thickness gastric resection | one week after surgery
  Success of the endoscopic resection will be defined by efficacy and safety: 1) Efficacy is defined as obtaining a full thickness resection and 2) Safety is defined as the absence of serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rajan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States